CLINICAL TRIAL: NCT03503162
Title: Evaluation of the Bowel Cleansing in Hospitalized Patients Using Pure-Vu System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL00044
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-10

CONDITIONS: Gastrointestinal Disease; Colorectal Cancer
Keywords: bowel prepartion
MeSH Terms: conditions — Gastrointestinal Diseases; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Colonoscopy with Pure-Vu System (Experimental): Standard colonoscopy procedure with Pure-Vu System
  Interventions: Device: Pure-Vu System

INTERVENTIONS:
Device: Pure-Vu System — The Pure-Vu System is FDA cleared device and CE marking received in February 2018, intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating or cleaning the colon and evacuating the irrigation fluid (water), feces and other bodily fluids and matter, e.g. blood.

SUMMARY:
The aim of this study is to evaluate the potential improvement in colonoscopy procedure's outcomes when using the Pure-Vu System in hospitalized patients who are indicated for colonoscopy procedure.

DETAILED DESCRIPTION:
This multi-center, prospective, single arm study will include up to 100 patients (20-40 patients per site), aimed at evaluating the performance of the Pure-Vu System in cleansing hospitalized patients' colon who are indicated for standard colonoscopy procedure.

Subjects will be enrolled at up to 4 clinical sites in the United States and Europe. Subjects who meet the eligibility criteria will be prescribed a standard bowel preparation bowel preparation regimen including diet restrictions and oral bowel preparation.

Following the bowel preparation, the patient will undergo colonoscopy with the Pure-Vu system.

In case of inadequate bowel preparation, as per the nurse report and / or BBPS < 2, in at least one of the colon segments, prior Pure-Vu use, the physician will complete a questionnaire on the patient's management standard of care assuming the absence of Pure-Vu.

Follow-up will be conducted at 48 hours (± 48 hours) post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients who are indicated for a screening, diagnostic, surveillance or therapeutic colonoscopy
2. Patients' age > 22 years
3. Patient has signed the informed consent

Exclusion Criteria:

1. Patients with known Inflammatory Bowel Disease and / or active Colitis
2. Patients with active diverticulitis
3. Patients with known or detected (during colonoscopy) bowel obstruction
4. Patients with BMI ≤ 18
5. Patients with ascites Child Pugh C
6. Patients who are 30 days post-transplant
7. Patients treated with Peritoneal dialysis
8. Patients under active IV inotropic medications
9. Patients with LVAD
10. Patients who have active anticoagulant medications (excluding aspirin) or dual antiplatelet therapy in their system prior to the procedure. (Note: to avoid exclusion therapy should be discontinued 48 hours or greater prior to the procedure based on discretion of physician)
11. Subjects with known coagulation disorder (INR ≥ 2 or platelets <50,000)
12. Subjects with hemodynamic instability.
13. Pregnancy (as stated by patient) or breast feeding
14. Subjects with altered mental status/inability to provide informed consent
15. Patients who have participated in another interventional clinical study in the last 2 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Choi, Study Director — Motus GI Technologies Ltd.
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
no plan to share the individual participated date with other researchers at this point.

REFERENCES:
- [Derived] Neumann H, Latorre M, Zimmerman T, Lang G, Samarasena J, Gross S, Brahmbhatt B, Pazwash H, Kushnir V. A multicenter, prospective, inpatient feasibility study to evaluate the use of an intra-colonoscopy cleansing device to optimize colon preparation in hospitalized patients: the REDUCE study. BMC Gastroenterol. 2021 May 22;21(1):232. doi: 10.1186/s12876-021-01817-2. PMID 34022813

RESULTS

PARTICIPANT FLOW:
Groups:
- Colonoscopy With Pure-Vu System: Inpatient colonoscopies with Pure-Vu System- Single Arm
  Pure-Vu System: The Pure-Vu System is FDA cleared device intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating or cleaning the colon and evacuating the irrigation fluid (water), feces and other bodily fluids and matter, e.g. blood.
Period: Overall Study
Arm/Group | Colonoscopy With Pure-Vu System
Started | 95
Completed | 94
Not Completed | 1
Not completed — did not meet eligibility | 1

BASELINE CHARACTERISTICS:
Arm/Group | Colonoscopy With Pure-Vu System
Number analyzed (Participants) | 94
Age, Customized [Mean (Full Range); unit: years] | 62.44 [28 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 69
  Germany | 25

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Adequate Cleansing Level Before and After the Use of the Pure-Vu System
Description: The rate of adequate cleansing level in each colon segment before and after use of Pure-Vu will be evaluated using the Boston Bowel Preparation Scale (BBPS). Segment score of 0-3 given to each of the 3 segments of the colon (Left side, Transverse and right side) summed for the maximum score of 9 (0= dirtiest and 9= pristine).
  An adequate cleansing procedure will be considered when all the colon segments will be graded as 2 or above.
Time Frame: up to 2 hours
Population: Rate of Adequacy of bowel preparation using the Boston Bowel Preparation Score (BBPS)
Measure: Mean (95% Confidence Interval); unit: Percentage of Adequate cleansing
Groups:
- Colonoscopy With Pure-Vu System: Inpatient colonoscopy procedure with Pure-Vu System
  Pure-Vu System: The Pure-Vu System is FDA cleared device and CE marking received in February 2018, intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating or cleaning the colon and evacuating the irrigation fluid (water), feces and other bodily fluids and matter, e.g. blood.
Arm/Group | Colonoscopy With Pure-Vu System
Number analyzed (Participants) | 84
Percentage of Adequate cleansing
  Rate of adequate preparation measured by BBPS before Pure-Vu Use | 38 [28 to 49]
  Rate of adequate preparation measured by BBPS after Pure-Vu Use | 96 [90 to 99]

ADVERSE EVENTS:
Time Frame: From procedure to 48 hours post procedure
Arm/Group | Colonoscopy With Pure-Vu System
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 1/94
Other Adverse Events (participants affected / at risk) | 3/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colonoscopy With Pure-Vu System (N=94)
Perforation (Gastrointestinal disorders) | 1 (1) — After procedure patient reported abdominal pain. Exploratory laparoscopy was performed and an 1 cm tear was repaired with suturing. Patient tolerated the procedure well and discharged 2 days post op. Event was related to retroflexion.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colonoscopy With Pure-Vu System (N=94)
Fever (Gastrointestinal disorders) | 1 (1) — Severity was Mild and resolved in 1 day.
abdominal pain (Gastrointestinal disorders) | 1 (1) — Severity was Mild and resolved in 1 day.
Drop in Hemoglobin (Gastrointestinal disorders) | 1 (1) — Severity was Mild and resolved in 2 day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT03503162/Prot_SAP_001.pdf